CLINICAL TRIAL: NCT06261762
Title: Hard and Soft Tissue Dimensional Change After Consecutive Extractions and Unassisted Socket Healing in the Esthetic Zone: A Pilot Study
Brief Title: Hard and Soft Tissue Dimensional Change After Consecutive Extractions and Unassisted Socket Healing in the Esthetic Zone
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Other Study IDs: SDC-24-1
Record Dates: First submitted 2024-02-07; First posted 2024-02-15 (Actual); Last update posted 2024-02-15 (Actual); Status verified 2024-02

CONDITIONS: Wound Heal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this observational study is to evaluate the post-extraction hard and soft tissue dimension changes in patients requiring consecutive extractions and unassisted socket healing in the anterior maxilla. The main questions it aims to answer are:

* Is significant alveolar ridge resorption observed at center sites after consecutive extractions
* Is significant alveolar ridge resorption observed at the interalveolar septum after consecutive extractions, are different extraction sites associated with significantly different bone resorption
* Is a thick or thin wall phenotype associated with the amount of bone resorption
* Is soft tissue thickness change associated with the corresponding location (extraction site or interalveolar septum) and post-extraction thickness of the bone
* Is the interdental papilla height significantly affected after extractions.

Participants will undergo consecutive (two) extractions and will be evaluated after subsequent unassisted socket healing for 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* Require consecutive (two) teeth replacement in the anterior maxilla
* Signed informed consent
* No significant medical conditions
* Patients with healthy periodontal conditions or previously treated to controlled and stable conditions

Exclusion Criteria:

* General medical (American Society of Anesthesiologists, ASA, class III or IV) and/or psychiatric contraindications
* Pregnancy or nursing
* Any interfering medication such as steroid therapy or bisphosphonate therapy
* Uncontrolled diabetes
* Autoimmune diseases or inflammatory diseases affecting the intraoral tissues
* Radiation therapy to head or neck region

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The group is selected from the referred patient pool. Age 18 or older. Absence of significant medical conditions. Sites with a need for consecutive (two) teeth extraction in the anterior maxilla.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-29 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Bone level change from baseline | Baseline and at 8 weeks
  Measured in millimeters using segmented surface model superimpositions. Changes in bone loss between baseline and an 8 week healing period using CBCT. From the Digital Imaging and Communications in Medicine (DICOM) files two surface mesh models were generated, which were superimposed and the changes were subsequently analyzed.
Soft tissue change from baseline | Baseline and at 8 weeks
  Changes in soft tissue loss at baseline and 8 weeks were analyzed using digital dental impressions acquired from intraoral scans, which were superimposed and the changes were analyzed.

SECONDARY OUTCOMES:
Correlation between baseline facial bone thickness and dimensional soft tissue alterations during healing at the interalveolar septum. | Baseline and at 8 weeks
  To measure correlation, the Spearman Rank Correlation Coefficient was calculated. Nonparametric models for longitudinal data were applied to analyze the impact of bone wall phenotype and healing period upon dimensional alterations.

CONTACTS AND LOCATIONS:
Overall Officials: Feng Wang, Principal Investigator — Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University